CLINICAL TRIAL: NCT04226560
Title: Clinical Evaluation of the Clinical Performance and Safety of a New Monthly Disposable Silicone Hydrogel Soft Contact Lenses
Brief Title: Performance and Safety of Silicone Hydrogel Soft Contact Lenses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ApexLens Co., Ltd. (Industry)
Collaborators: Chang Gung Memorial Hospital (Other); Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ApexLens-201901
Record Dates: First submitted 2020-01-02; First posted 2020-01-13 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Myopia
Keywords: Nearsightedness; Eye wear; Myopia control; Contact lens
MeSH Terms: conditions — Myopia | interventions — Contact Lenses; Hydrophobic and Hydrophilic Interactions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 41% Silicone hydrogel Soft contact lenses (SHSCL) (Experimental): Healthy adult males or females age ≥20-45 years of age
  Interventions: Device: 41% Silicone Hydrogel Soft Contact Lenses(SHSCL); Other: Contact Lens Care Product; Other: Contact Lens Case
- ACUVUE® VITA™ (Active Comparator): Healthy adult males or females age ≥20-45 years of age
  Interventions: Device: ACUVUE® VITA™ (senofilcon C) Brand (Soft) Contact Lens; Other: Contact Lens Care Product; Other: Contact Lens Case

INTERVENTIONS:
Device: 41% Silicone Hydrogel Soft Contact Lenses(SHSCL) — Silicone Hydrogel
  Arms: 41% Silicone hydrogel Soft contact lenses (SHSCL)
Device: ACUVUE® VITA™ (senofilcon C) Brand (Soft) Contact Lens — Senofilcon C (USFDA Device License #K160212)
  Arms: ACUVUE® VITA™
Other: Contact Lens Care Product — Cefatrizine (propylene Glycol), Sodium Citrate (sodium Citrate Tribasic), Sodium Chloride, Sodium Borate (sodium Biboratesodium Tetraborate, Polyquaternium -1, Hydrochloric Acid, Sodium Hydroxide, Water Purified ( Eq to Aqueous Purified Or Purified Water ), Tetronic 1304, Myristamidopropyl Dimethylamine, Nonanoyl Ethylenediaminetriacetic Acid
  Other Names: Opti-Free Replenish Multi-purpose Disinfecting Solution
Other: Contact Lens Case — "Alcon" Soft (hydrophilic) Contact Lens Case (Non-Sterile)
  Other Names: "Alcon" Soft (hydrophilic) Contact Lens Case (Non-Sterile)

SUMMARY:
To demonstrate substantial equivalence of the new Silicone Hydrogel Soft Contact Lenses(SHSCL) to the commercially available ACUVUE® VITA™ contact lens

DETAILED DESCRIPTION:
This study is a prospective, subject-masked, bilateral, randomized, parallel group dispensing study comparing the SHSCL test lens against the 1-Month ACUVUE® VITA™ (1-MAV) control lenses. Each subject will be randomized to wear either the test or of the control with similar/comparable lens parameters optimized for vision.

Both test and control lens will be used in their daily wear, monthly replacement modality for thirteen (13) weeks. It is anticipated that this study will involve up to 6 scheduled visits.

ELIGIBILITY:
Inclusion Criteria:

A person is eligible for inclusion in the study if he/she:

1. Healthy adult males or females age ≥20-45 years of age;
2. Be a currently adapted soft contact lens wearer (i.e. be wearing lenses at least 1 month prior to enrolment) and the last contact lenses worn more than a week ago;
3. Have a contact lens powers between -2.00D and -6.00D (both inclusive) in both eyes;
4. Astigmatism of 1.00D or less in both eyes;
5. Be able to wear the lens powers available for this study;
6. Be correctable to a visual acuity of 0.8 decimal (+0.10 logMAR) or better in each eye;
7. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol;
8. The subject must read and sign the Informed Consent form.

Exclusion Criteria:

A person will be excluded from the study if he/she:

1. Previously unsuccessful with contact lens wear, worn rigid gas permeable contact lenses within past 12 months;
2. Women who are pregnant, lactating or planning a pregnancy at the time of enrolment (by verbal confirmation at the screening visit);
3. Any ocular or systemic allergies or diseases that may contraindicate contact lens wear;
4. Any ocular medications use within the last one month;
5. Any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear;
6. Any infectious disease (e.g., hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g., HIV), by self-report;
7. Any current or previous orthokeratology treatment, or planned for orthokeratology treatment during the study;
8. Any previous history of ocular and/or refractive surgery (e.g., radial keratotomy, PRK, LASIK, etc.), or planned for ocular and/or refractive surgery during the study
9. History of herpetic keratitis;
10. History of binocular vision abnormality or strabismus, by self-report;
11. Allergic reactions to test lens, control lens or the contact lens solution used in this study;
12. A clinical finding or history of entropion, ectropion, chalazia, recurrent styes, glaucoma, pathologically dry eye, history of recurrent corneal erosions, aphakia, or moderate or above corneal distortion, by self-report;
13. Employee of investigational clinic (e.g., Investigator, Coordinator, Technician);
14. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment;
15. Any slit lamp findings which would contraindicate contact lens wear;
16. Any history of a contact lens-related corneal inflammatory event within the past 12 months that may contraindicate contact lens wear; or
17. Clinically significant (grade 3 or 4) anterior segment abnormalities or any infection of the eye, lids, or associated structures;
18. Subjects are considered ineligible for the study as judged by the investigator.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Estimated)
Dates: Start 2020-04-20 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Best-corrected contact lens visual acuity | 13 weeks
  The primary efficacy endpoint in this evaluation is the percentage of subjects with best-corrected contact lens visual acuity of 0.8 decimal (+0.10 logMAR) and 1.0 decimal (0.00 logMAR) or better.
  The Snellen chart will be used for visual acuity testing.
Permanent loss of visual acuity | 13 weeks
  The primary safety endpoint in this evaluation is the percentage of subjects with permanent loss of two or more lines of visual acuity.
Serious adverse reactions | 13 weeks
  The primary safety endpoint in this evaluation is the rate of serious adverse reactions related to visual acuity loss as well as accompanying slit-lamp findings and other associated observations.

SECONDARY OUTCOMES:
Lens comfort | 13 weeks
  The secondary efficacy endpoint is the assessment of lens comfort over time with the lens for the recommended wearing time. This will be measured using Study Diary.
  Subject will be given a Study Diary to be completed at home, to reflect their lens wear experience at the time of rating. Subject will be given careful explanation of how and when to complete them.
  Comfort after insertion (i.e. after lens settling), after 4 hours, and just before lens removal (0-10 scale)(10 = cannot be felt, 0 = painful)
Symptoms of dryness | 13 weeks
  The secondary efficacy endpoint is the assessment of dryness symptoms with the lens for the recommended wearing time. This will be measured using Study Diary.
  Subject will be given a Study Diary to be completed at home, to reflect their lens wear experience at the time of rating. Subject will be given careful explanation of how and when to complete them.
  Dryness after insertion (i.e. after lens settling), after 4 hours, and just before lens removal (0-10 scale)(10 = cannot be felt, 0 = painful)
Slit lamp findings | 13 weeks
  The secondary efficacy endpoint is the assessment of the rate of any Slit Lamp Findings > Grade 2.
  The subject will be instructed to take off the study lenses before the slit-lamp biomicroscopy assessment.
  Slit-lamp biomicroscopy will be assessed according to the approved study biomicroscopy CRF.
  ISO 11980:2012 Annex B will be used to grade the Slit-lamp findings.
Subject reported ocular complaints | 13 weeks
  Subjects will be asked to assess ocular complaints by using Study Diary.

CONTACTS AND LOCATIONS:
Overall Officials: Yih-Shiou Hwang, M.D.,Ph.D., Principal Investigator — Chang Gung Memorial Hospital; Hsin-Wei Huang, M.D., Principal Investigator — Taipei Medical University - Municipal Wan Fang Hospital
Locations (1):
- ApexLens Co., Ltd., Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dumbleton KA, Woods CA, Jones LW, Fonn D. The relationship between compliance with lens replacement and contact lens-related problems in silicone hydrogel wearers. Cont Lens Anterior Eye. 2011 Oct;34(5):216-22. doi: 10.1016/j.clae.2011.03.001. Epub 2011 Apr 13. PMID 21493121